CLINICAL TRIAL: NCT06755736
Title: The Effect of Superficial Cervical Block Application on Postoperative Opioid Consumption in Patients Undergoing Anterior Cervical Discectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-10840098-202.3.02-7384
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Superficial Cervical Block; Postoperative Pain
Keywords: superficial cervical block; anterior cervical discectomy; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): 1 g intravenous paracetamol and 100 mg intravenous tramadol will be administered 30 minutes before the end of surgery. In addition, 4 mg intravenous ondansetron will be given to prevent postoperative nausea and vomiting.
- superficial cervical block (Experimental): In addition to routine analgesics applied to the control group, a superficial cervical block will be applied immediately before awakening. The block is performed with the patient in the supine position. A high-frequency (11-12 MHz) linear ultrasound probe is placed at the midpoint of the sternocleidomastoid (SCM) muscle. The ultrasound probe is placed in the transverse plane. During the block, the needle is monitored on the ultrasound image using the in-plane technique. The needle is advanced caudally and directed under the sternocleidomastoid muscle, just above the prevertebral fascia. : The correct position of the needle is confirmed under ultrasound guidance. First, 1-2 ml of saline is injected to confirm the correct location. Then, 20 ml of 0.25% bupivacaine local anesthetic is applied behind the sternocleidomastoid muscle between the muscle and the prevertebral fascia.
  Interventions: Drug: superficial cervical plexus block

INTERVENTIONS:
Drug: superficial cervical plexus block — In anterior cervical discectomy surgeries, superficial cervical block will be used for analgesia.
  Arms: superficial cervical block

SUMMARY:
This randomized controlled trial aims to evaluate the effect of superficial cervical block on postoperative opioid consumption in patients undergoing anterior cervical discectomy surgery. Postoperative pain significantly impacts recovery and patient comfort in this type of surgery, where symptoms such as swallowing difficulties, occipito-cervical pain, and positional discomfort are common. While opioids are effective for pain control, their side effects, such as nausea, vomiting, and respiratory depression, may lead to complications, especially in cervical surgeries with potential airway risks.

Superficial cervical block is a simple and safe regional anesthesia technique proven effective in managing pain after thyroid and carotid surgeries. However, its potential benefits in anterior cervical discectomy surgeries have not been extensively studied.

Our hypothesis is that superficial cervical block can reduce postoperative opioid use and provide effective pain management for these patients. Additionally, investigators aim to compare opioid-related side effects and postoperative pain scores between groups with and without the block.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial will be conducted at Medipol Mega University Hospital on patients undergoing anterior cervical discectomy surgery. The study's primary objective is to assess the impact of superficial cervical block on postoperative opioid consumption. Secondary objectives include comparing opioid-related side effects, such as nausea, vomiting, and respiratory depression, and evaluating patients' postoperative Numerical Rating Scale (NRS) pain scores.

Patient Selection:

Eligible participants are aged 18-80 years, with an American Society of Anesthesiologists (ASA) physical status of I-III. Patients with allergies, pregnancy, or neurological/psychiatric conditions will be excluded.

Study Groups:

Participants will be randomly assigned to two groups:

Group 1 (Control): No block will be administered. Group 2 (Intervention): A superficial cervical block will be performed before waking the patient.

Anesthesia Management:

All patients will receive a standard anesthesia protocol, including midazolam, propofol, fentanyl, and rocuronium for induction, followed by maintenance with oxygen-air mix and additional doses of midazolam, fentanyl, and rocuronium. Postoperatively, 1 g paracetamol and 100 mg tramadol will be administered, along with ondansetron to prevent nausea.

Block Technique:

In Group 2, the superficial cervical block will be performed after the surgery is completed but before the patient is awakened. Under sterile conditions and ultrasound guidance, 20 mL of 0.25% bupivacaine will be injected near the superficial branches of the cervical nerves.

Postoperative Evaluation:

Patients' pain levels will be assessed using the Numerical Rating Scale (NRS) at specific intervals (recovery, 3, 6, 12, 18, and 24 hours). A rescue analgesic (1 mg/kg tramadol) will be provided if the NRS score is ≥4. Postoperative opioid consumption, side effects, and complications, including nausea, vomiting, itching, and block-related hematomas, will be recorded.

This study aims to provide valuable insights into the role of superficial cervical block in improving pain management and reducing opioid-related risks in anterior cervical discectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for anterior cervical discectomy surgery
* aged between 18 and 80 years,
* American Society of Anesthesiology (ASA) physical status I-III, scheduled for anterior cervical discectomy surgery will be included.

Exclusion Criteria:

* history of allergies,
* allergic to local anesthetics,
* pregnant women
* psychiatric or neurological disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of superficial cervical block application on postoperative opioid use in patients undergoing cervical discectomy surgery via anterior approach. | first 24 hours after the operation
  The amount of tramadol used as rescue analgesic will be compared between the groups.

SECONDARY OUTCOMES:
The aim of this study is to compare postoperative NRS (Numerical Rating Scale) pain scores of the patients between the groups. | first 24 hours after the operation
  The NRS is an 11-point scale. Zero means 'no pain', 10 means 'the most severe pain imaginable'. NRS scores at rest and during mobilization are evaluated and recorded in the postoperative recovery unit at 3, 6, 12, 18 and 24 hours. If the NRS score is ≥ 4, 1 mg kg-1 IV tramadol is administered as a rescue analgesic.

OTHER OUTCOMES:
The aim of this study is to compare opioid-related side effects (such as nausea, vomiting, respiratory depression) of the patients between the groups. | first 24 hours after the operation
  It will be evaluated whether there are any opioid-related side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Ömür, Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication

REFERENCES:
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Elvir-Lazo OL, White PF. The role of multimodal analgesia in pain management after ambulatory surgery. Curr Opin Anaesthesiol. 2010 Dec;23(6):697-703. doi: 10.1097/ACO.0b013e32833fad0a. PMID 20847690
- [Background] Mariappan R, Mehta J, Massicotte E, Nagappa M, Manninen P, Venkatraghavan L. Effect of superficial cervical plexus block on postoperative quality of recovery after anterior cervical discectomy and fusion: a randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):883-90. doi: 10.1007/s12630-015-0382-3. Epub 2015 Apr 14. PMID 25869024